CLINICAL TRIAL: NCT01172938
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Efficacy and Safety Study of Two Doses of Apremilast (CC-10004) in Subjects With Active Psoriatic Arthritis
Brief Title: Efficacy and Safety Study of Apremilast to Treat Active Psoriatic Arthritis
Acronym: PALACE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSA-002
Record Dates: First submitted 2010-07-06; First posted 2010-07-30 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Psoriasis; Arthritis; inflammation; skin condition; inflammatory cells; apremilast; CC-10004; phosphodiesterase type 4
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Arthritis; Inflammation; Skin Diseases | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Apremilast 20 mg (Experimental): 20 mg Apremilast tablets administered twice daily for 24 weeks during the placebo-controlled phase followed by 20 mg Apremilast tablets administered twice daily for up to 4.5 years in the active treatment / long-term safety phase
  Interventions: Drug: Apremilast 20mg
- Apremilast 30mg (Experimental): 30 mg Apremilast tablets administered twice a day for 24 weeks during the placebo-controlled phase followed by 30 mg Apremilast tablets administered twice a day for up to 4.5 years in the active treatment / long-term safety phase orally twice daily
  Interventions: Drug: Apremilast 30mg
- Placebo + 20 mg Apremilast (Placebo Comparator): Placebo + 20 mg Apremilast tablets administered twice daily for 24 weeks during the placebo-controlled phase followed by 20 mg Apremilast tablets administered twice daily for up to 4.5 years in the active treatment / long-term safety phase. Subjects who do not have at least 20% improvement in their swollen and tender joint counts at Week 16 will escape to 20 mg Apremilast twice daily at Week 16
  Interventions: Drug: Placebo + 20 mg Apremilast
- Placebo + 30 mg Apremilast (Placebo Comparator): Placebo + 30 mg Apremilast tablets administered twice daily for 24 weeks during the placebo-controlled phase followed by 30 mg Apremilast tablets administered twice daily for up to 4.5 years in the active treatment / long-term safety phase. Subjects who do not have at least 20% improvement in their swollen and tender joint counts at Week 16 will escape to 30 mg Apremilast twice daily at Week 16.
  Interventions: Drug: Placebo + 30 mg Apremilast

INTERVENTIONS:
Drug: Apremilast 20mg — Apremilast 20 mg twice daily, orally
  Other Names: CC-10004
  Arms: Apremilast 20 mg
Drug: Apremilast 30mg — Apremilast 30 mg twice daily, orally
  Other Names: CC-10004
  Arms: Apremilast 30mg
Drug: Placebo + 20 mg Apremilast — Placebo + 20 mg Apremilast
  Other Names: Placebo; CC-10004
  Arms: Placebo + 20 mg Apremilast
Drug: Placebo + 30 mg Apremilast — Placebo + 30 mg Apremilast
  Other Names: Placebo; CC-10004
  Arms: Placebo + 30 mg Apremilast

SUMMARY:
The purpose of this study is to determine whether apremilast is safe and effective in the treatment of patients with psoriatic arthritis, specifically in improving signs and symptoms of psoriatic arthritis (tender and swollen joints, pain, physical function) in treated patients.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is an inflammatory arthritis that occurs in 6-39% of psoriasis patients. The immunopathogenesis of PsA, which mirrors but is not identical to that seen in psoriatic plaques, reflects a complex interaction among resident dendritic, fibroblastic and endothelial cells, and inflammatory cells attracted to the synovium by cytokines and chemokines. Apremilast (CC-10004) is a novel oral agent that modulates multiple inflammatory pathways through targeted phosphodiesterase type 4 (PDE4) enzyme inhibition. Therefore, apremilast has the potential to be effective in the treatment of PsA.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged ≥ 18 years at time of consent.
* Have a diagnosis of Psoriatic Arthritis (PSA, by any criteria) of ≥ 6 months duration.
* Meet the Classification Criteria for Psoriatic Arthritis (CASPAR) at time of screening.
* Must have been inadequately treated by disease-modifying antirheumatic drugs (DMARDs)
* May not have axial involvement alone
* Concurrent treatment allowed with methotrexate, leflunomide, or sulfasalazine
* Have ≥ 3 swollen AND ≥ 3 tender joints.
* Males & Females must use contraception
* Stable dose of nonsteroidal anti-inflammatory drugs (NSAIDs), narcotics and low dose oral corticosteroids allowed.

Exclusion Criteria:

* Pregnant or breast feeding.
* History of allergy to any component of the investigational product.
* Hepatitis B surface antigen and/or Hepatitis C antibody positive at screening.
* Therapeutic failure on > 3 agents for PsA or > 1 biologic tumor necrosis factor (TNF) blocker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2010-06-02 (Actual); Primary Completion 2012-04-27 (Actual); Study Completion 2016-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (92):
- United States (27):
  - Achieve Clinical Research LLC, Birmingham, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - UCSD-Thornton Hospital, La Jolla, California
  - Stanford University Medical Center, Palo Alto, California
  - Inland Rheumatology Clinical Trials, Upland, California
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - North Florida Dermatology, Jacksonville, Florida
  - Tampa Medical Group Pa, Tampa, Florida
  - Sonora Clinical Research, LLC, Boise, Idaho
  - Coeur D'Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - The Arthritis Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers, Michigan City, Indiana
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Justus Fiechtner MD PC, Lansing, Michigan
  - Physicians East, Greenville, North Carolina
  - Carolina Bone and Joint, Monroe, North Carolina
  - Piedmont Medical Research Associates Inc, Winston-Salem, North Carolina
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, LLP, West Reading, Pennsylvania
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Accurate Clinical Research Inc, Houston, Texas
  - Arthritis and Osteoporosis Associates LLP, Lubbock, Texas
  - Center for Clinical Studies, Webster, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Rheumatology Associates, Seattle, Washington
  - Arthritis Northwest Rheumatology, Spokane, Washington
- Australia (5):
  - Monash Medical Centre, Clayton, Victoria
  - Eastern Health Clinical School, Box Hill
  - Repatriation General Hospital, Daws Park
  - St Vincent's Hospital Melbourne, Fitzroy
  - Emeritus Research, Malvern
- Austria (3):
  - Ordination Wien Dr. Hanusch, Vienna
  - Medizinische Universitat Wien, Vienna
  - Kaiser-Franz-Josef Spital, Vienna
- Canada (16):
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - St. Clare's Health Care Corporation of St. John's, St. John's, Newfoundland and Labrador
  - Ultranova Skincare, Barrie, Ontario
  - MAC Research Incorporated, Hamilton, Ontario
  - K-W Musculoskeletal Research Inc., Kitchener, Ontario
  - Saint Josephs Healthcare System, London, Ontario
  - Credit Valley Professional Building, Mississauga, Ontario
  - The Arthritis Program Research Group Inc., Newmarket, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Probity Medical Research Inc, Waterloo, Ontario
  - Jude Rodrigues Private Practice, Windsor, Ontario
  - Hospital Maisonneuve - Rosemont, Montreal, Quebec
  - Institut de Rhumatologie de Montreal, Montreal, Quebec
  - Centre de Rhumatologie St-Louis, Sainte-Foy, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Hospital Fleurimont, Sherbrooke, Quebec
  - Saskatoon Osteoporosis Centre, Saskatoon, Saskatchewan
- France (2):
  - Ipros - Chr Orleans, Orléans
  - Hopital Purpan, Toulouse
- Germany (5):
  - Klinikum Duisburg, Wedau Kliniken, Duisburg
  - Friedrich-Alexander-Universiät Erlangen Nürnberg, Erlangen
  - Allgemeines Krankenhaus Eilbeck, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - Praxis Prof. Herbert Kellner, München
- Hungary (5):
  - Qualiclinic kft, Budapest
  - Synexus Magyarország Kft., Budapest
  - Honvéd Kórház - Állami Egészségügyi Központ, Budapest
  - MAV Korhaz es Rendelointezet Szolnok, Szolnok
  - Veszprém Megyei Önkormányzat Csolnoky Ferenc Kórház-Rendelöintézet, Veszprém
- New Zealand (6):
  - P3 Research, Crofton Downs
  - Waikato hospital, Hamilton
  - Middlemore Clinical Trials, New Zealand
  - Queen Elizabeth Hospital for Rheumatic Disease, Rotorua
  - North Shore Hospital, Takapuna
  - Timaru Hospital, Timaru
- Poland (6):
  - Szpital Uniwersytecki im. Dr A.Jurasza, Bydgoszcz
  - Szpital Uniwersytecki nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Synexus SCM Sp. z o.o., Gdynia
  - Synexus SCM Sp. z o.o., Katowice
  - Wojewodzki Zespol Reumatologiczny, Sopot
  - Synexus SCM Sp. z o.o. Oddz. Warszawa, Warsaw
- Russia (5):
  - Kemerovo State Medical Academy, Kemerovo
  - Ryazan I.P. Pavlov State Medical University, Ryazan
  - Departmental Hospital at Smolensk Station RZhD JSC, Smolensk
  - Regional Clinical Hospital, Vladimir
  - Voronezh Regional Clinical Hopsital #1, Voronezh State Medical Academy, Voronezh
- South Africa (5):
  - Panorama Medical Centre, Cape Town
  - Groote Schuur Hospital, Cape Town
  - Chelmsford Medical Centre 2, Durban
  - Clinresco Centres Pty Ltd, Johannesburg
  - The Park, Pinelands
- Spain (4):
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
- United Kingdom (3):
  - Barnsley Hospital, Barnsley South Yorkshire
  - Colchester General Hospital, Colchester
  - West Suffolk Hospital, Edmunds

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Result] Kavanaugh A, Mease PJ, Gomez-Reino JJ, Adebajo AO, Wollenhaupt J, Gladman DD, Hochfeld M, Teng LL, Schett G, Lespessailles E, Hall S. Longterm (52-week) results of a phase III randomized, controlled trial of apremilast in patients with psoriatic arthritis. J Rheumatol. 2015 Mar;42(3):479-88. doi: 10.3899/jrheum.140647. Epub 2015 Jan 15. PMID 25593233
- [Derived] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690
- [Derived] Mease PJ, Gladman DD, Kavanaugh A, McGonagle D, Nash P, Guerette B, Nakasato P, Brunori M, Teng L, McInnes IB. Articular and Extra-Articular Benefits in ACR20 Non-responders at Week 104 Treated With Apremilast: Pooled Analysis of Three Randomized Controlled Trials. Rheumatol Ther. 2021 Dec;8(4):1677-1691. doi: 10.1007/s40744-021-00369-x. Epub 2021 Sep 18. PMID 34536218
- [Derived] Mease PJ, Gladman DD, Ogdie A, Coates LC, Behrens F, Kavanaugh A, McInnes I, Queiro R, Guerette B, Brunori M, Teng L, Smolen JS. Treatment-to-Target With Apremilast in Psoriatic Arthritis: The Probability of Achieving Targets and Comprehensive Control of Disease Manifestations. Arthritis Care Res (Hoboken). 2020 Jun;72(6):814-821. doi: 10.1002/acr.24134. Epub 2020 May 8. PMID 31909868
- [Derived] Kavanaugh A, Gladman DD, Edwards CJ, Schett G, Guerette B, Delev N, Teng L, Paris M, Mease PJ. Long-term experience with apremilast in patients with psoriatic arthritis: 5-year results from a PALACE 1-3 pooled analysis. Arthritis Res Ther. 2019 May 10;21(1):118. doi: 10.1186/s13075-019-1901-3. PMID 31077258
- [Derived] Gladman DD, Kavanaugh A, Gomez-Reino JJ, Wollenhaupt J, Cutolo M, Schett G, Lespessailles E, Guerette B, Delev N, Teng L, Edwards CJ, Birbara CA, Mease PJ. Therapeutic benefit of apremilast on enthesitis and dactylitis in patients with psoriatic arthritis: a pooled analysis of the PALACE 1-3 studies. RMD Open. 2018 Jun 27;4(1):e000669. doi: 10.1136/rmdopen-2018-000669. eCollection 2018. PMID 30018799
- [Derived] Kavanaugh A, Mease PJ, Gomez-Reino JJ, Adebajo AO, Wollenhaupt J, Gladman DD, Lespessailles E, Hall S, Hochfeld M, Hu C, Hough D, Stevens RM, Schett G. Treatment of psoriatic arthritis in a phase 3 randomised, placebo-controlled trial with apremilast, an oral phosphodiesterase 4 inhibitor. Ann Rheum Dis. 2014 Jun;73(6):1020-6. doi: 10.1136/annrheumdis-2013-205056. Epub 2014 Mar 4. PMID 24595547

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a multicenter study with 83 study sites from the US, Canada, Europe, Russia, Australia, New Zealand and South Africa.
Pre-assignment Details: The study population was restricted to male and female subjects ≥ 18 years of age with moderate to severe Psoriatic Arthritis (PsA). Participants must have had a diagnosis of PsA by the Classification Criteria for Psoriatic Arthritis (CASPAR) criteria, including peripheral joint involvement.
Groups:
- Placebo: Participants initially randomized to receive placebo tablets twice daily in the 24-week placebo-controlled phase. Participants who did not have at least 20% improvement in swollen and tender joint counts at Week 16 were re-randomized to either 20 mg or 30 mg apremilast twice daily (early escape).
- Apremilast 20 mg: Participants initially randomized to 20 mg apremilast tablets twice daily (BID) in the placebo-controlled phase and continued to receive 20 mg apremilast tablets BID in the active treatment / long-term safety phase. After 30 mg apremilast BID was identified as the optimal dose, all active subjects originally receiving 20 mg apremilast BID were switched to the 30 mg apremilast BID dose
- Apremilast 30 mg: Participants initially randomized to 30 mg apremilast tablets twice daily (BID) in the placebo-controlled phase and continued to receive 30 mg apremilast tablets BID for up to 4.5 years in the active treatment / long-term safety phase
- Placebo / Apremilast 20 mg EE: Participants initially randomized to receive placebo twice daily who were re-randomized due to early escape (EE) at Week 16 to receive 20 mg apremilast for up to 4.5 years. After 30 mg apremilast BID was identified as the optimal dose, all active participants originally receiving 20 mg apremilast BID were switched to the 30 mg apremilast BID dose for these participants.
- Placebo / Apremilast 20 mg XO: Participants initially randomized to receive placebo twice daily who were re-randomized at Week 24 (XO) to receive 20 mg apremilast for up to 4.5 years. After 30 mg apremilast BID was identified as the optimal dose, all active participants originally receiving 20 mg apremilast BID were switched to the 30 mg apremilast BID dose for these participants.
- Placebo / Apremilast 30 mg EE: Participants initially randomized to receive placebo twice daily who were re-randomized due to early escape (EE) at Week 16 to receive 30 mg apremilast for up to 4.5 years.
- Placebo / Apremilast 30 mg XO: Participants initially randomized to receive placebo twice daily who were re-randomized at Week 24 to receive 30 mg apremilast for up to 4.5 years.
- Placebo/Apremilast 20 mg (Long-Term Extension): Participants initially randomized to placebo tablets BID during the placebo controlled phase and were re-randomized to apremilast at Week 16 or Week 24 and continued receiving apremilast 20 mg BID for up to 4.5 years in the active treatment / long-term safety phase. After 30 mg apremilast BID was identified as the optimal dose, all active participants originally receiving 20 mg apremilast BID were switched to the 30 mg apremilast BID dose.
- Placebo/Apremilast 30 mg (Long-Term Extension): Participants initially randomized to placebo tablets BID during the placebo controlled phase and were re-randomized to apremilast 30 mg tablets BID at Week 16 or Week 24 and continued receiving apremilast 30 mg BID for up to 4.5 years in the active treatment / long-term safety phase.
Period: Placebo-controlled Phase (Week 0-24)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Extension) | Placebo/Apremilast 30 mg (Long-Term Extension)
Started | 168 | 168 | 168 | 0 | 0 | 0 | 0 | 0 | 0
Received Treatment | 168 | 168 | 168 | 0 | 0 | 0 | 0 | 0 | 0
Completed Week 16 | 158 | 158 | 154 | 0 | 0 | 0 | 0 | 0 | 0
Early Escape at Week 16 | 107 (Five participants who escaped early did not complete Week 24) | 78 (Six participants who escaped early did not complete Week 24) | 58 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 150 (One participant who completed Week 24 did not enter the active treatment phase) | 146 | 148 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 18 | 22 | 20 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 11 | 8 | 10 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Active Treatment Phase (Weeks 25-52)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Extension) | Placebo/Apremilast 30 mg (Long-Term Extension)
Started | 0 | 136 (Ten participants who completed Week 24 did not enter the active treatment phase) | 145 (Three participants who completed Week 24 did not enter the active treatment phase) | 51 (One participant who escaped early and completed Week 24 did not enter the active treatment phase) | 23 | 49 (One participant who escaped early and completed Week 24 did not enter the active treatment phase) | 24 | 0 | 0
Completed | 0 | 124 | 130 | 44 | 19 | 34 | 22 | 0 | 0
Not Completed | 0 | 12 | 15 | 7 | 4 | 15 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 5 | 1 | 1 | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 4 | 7 | 3 | 1 | 3 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 5 | 1 | 2 | 2 | 9 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Period: Active-Treatment Phase (Weeks 52-104)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Extension) | Placebo/Apremilast 30 mg (Long-Term Extension)
Started | 0 | 118 (Six participants who completed Week 52 did not enter the next year of active treatment phase) | 121 (Nine participants who completed Week 52 did not enter the next year of active treatment phase) | 0 | 0 | 0 | 0 | 61 | 49
Completed | 0 | 95 | 100 | 0 | 0 | 0 | 0 | 46 | 45
Not Completed | 0 | 23 | 21 | 0 | 0 | 0 | 0 | 15 | 4
Not completed — Adverse Event | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Lack of Efficacy | 0 | 7 | 8 | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Non-compliance with Study Drug | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 10 | 8 | 0 | 0 | 0 | 0 | 5 | 2
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Miscellaneous | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Missing | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Active-Treatment Phase Weeks (104-156)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Extension) | Placebo/Apremilast 30 mg (Long-Term Extension)
Started | 0 | 95 | 100 | 0 | 0 | 0 | 0 | 46 | 45
Completed | 0 | 84 | 93 | 0 | 0 | 0 | 0 | 41 | 41
Not Completed | 0 | 11 | 7 | 0 | 0 | 0 | 0 | 5 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 6 | 3 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Miscellaneious | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Active-Treatment Phase (Weeks 156-208)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Extension) | Placebo/Apremilast 30 mg (Long-Term Extension)
Started | 0 | 84 | 93 | 0 | 0 | 0 | 0 | 41 | 41
Completed | 0 | 75 | 88 | 0 | 0 | 0 | 0 | 32 | 34
Not Completed | 0 | 9 | 5 | 0 | 0 | 0 | 0 | 9 | 7
Not completed — Adverse Event | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 2 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Active-Treatment Phase (Weeks 208-260)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Extension) | Placebo/Apremilast 30 mg (Long-Term Extension)
Started | 0 | 75 | 88 | 0 | 0 | 0 | 0 | 32 | 34
Switched From 20 mg to 30 mg BID | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 0
Completed | 0 | 72 | 80 | 0 | 0 | 0 | 0 | 29 | 32
Not Completed | 0 | 3 | 8 | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study drug | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set consisting of all participants who were randomized as specified in the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Total
Number analyzed (Participants) | 168 | 168 | 168 | 504
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (12.13) | 48.7 (10.99) | 51.4 (11.72) | 50.4 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 83 | 92 | 255
  Male | 88 | 85 | 76 | 249
Duration of psoriatic arthritis [Mean (Standard Deviation); unit: years] | 7.31 (7.118) | 7.18 (6.842) | 8.09 (8.092) | 7.53 (7.366)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 16
Description: Percentage of participants with an American College of Rheumatology 20% (ACR20) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 20% improvement in 78 tender joint count; • ≥ 20% improvement in 76 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-Reactive Protein.
Time Frame: Baseline and Week 16
Population: Full analysis set consisting of all participants randomized as specified in the protocol. Participants who withdrew early or who did not have sufficient data for a definitive determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 168 | 168 | 168
percentage of participants | 19.0 | 30.4 | 38.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; In order to maintain the Type 1 error at the 0.05 significance level, the Hochberg procedure was to be used. The results of the endpoint were to be considered statistically significant if both the 30 mg apremilast dose versus placebo comparison and the 20 mg versus placebo comparison were statistically significant at the 0.05 significance level, or one of the comparisons was statistically significant at the 0.025 level; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; 2-sided p-value is based on the Cochran-Mantel-Haenszel (CMH) test adjusting for baseline disease modifying antirheumatic drug (DMARD) use; Adjusted Difference = 19.0, 95% CI 2-sided [9.7 to 28.3] — Adjusted difference is the weighted average of the treatment differences across the 2 strata of baseline DMARD use with the CMH weights. The 2-sided 95% confidence interval (CI) is based on a normal approximation to the weighted average
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0166, Cochran-Mantel-Haenszel; 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 11.3, 95% CI 2-sided [2.2 to 20.4] — Adjusted difference is the weighted average of the treatment differences across the 2 strata of baseline DMARD use with the CMH weights. The 2-sided 95% CI is based on a normal approximation to the weighted average

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire- Disability Index (HAQ-DI) at Week 16
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire consisting of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from Baseline in the overall score indicate improvement in functional ability.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 16 are included; Last observation carried forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 165 | 163 | 159
units on a scale | -0.086 (0.0360) | -0.198 (0.0364) | -0.244 (0.0364)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Pairwise comparisons (30 mg vs placebo and 20 mg vs placebo) were conducted conditional on the primary endpoint results. If the primary endpoint was statistically significant for both apremilast dose groups, pairwise comparisons for the HAQ-DI were to be evaluated at the 0.05 level using the Hochberg procedure. If only one apremilast dose was statistically significant, then only the comparison between that apremilast dose and placebo was conducted for the HAQ-DI score, at the 0.025 level; Test type: Superiority or Other; p = 0.0017, ANCOVA; Based on an ANCOVA model with treatment group and baseline DMARD use as factors, and the baseline value as a covariate; LS Mean Difference = -0.159, 95% CI 2-sided [-0.258 to -0.060]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0252, ANCOVA; Based on an analysis of covariance (ANCOVA) model with treatment group and baseline DMARD use as factors, and the baseline value as a covariate; LS Mean Difference = -0.113, 95% CI 2-sided [-0.211 to -0.014]

3. Secondary Outcome: Percentage of Participants With an ACR 20 Response at Week 24
Description: Percentage of participants with an American College of Rheumatology 20% (ACR20) response at Week 24. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 20% improvement in 78 tender joint count; • ≥ 20% improvement in 76 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-Reactive Protein.
Time Frame: Baseline and Week 24
Population: Full analysis set; Participants who discontinued early, escaped early at Week 16 or who did not have sufficient data for a definitive determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 168 | 168 | 168
percentage of participants | 13.1 | 25.6 | 35.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Secondary endpoints from the placebo-controlled period (Weeks 16 and 24) were analyzed in a hierarchical fashion to control the Type I error rate as described above; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 22.2, 95% CI 2-sided [13.4 to 30.9] — Adjusted difference is the weighted average of the treatment differences across the 2 strata of baseline DMARD use with the Cochran-Mantel-Haenszel (CMH) weights. The 2-sided 95% CI is based on a normal approximation to the weighted average
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.0038, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 12.4, 95% CI 2-sided [4.2 to 20.7] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire- Disability Index (HAQ-DI) at Week 24
Description: as for outcome 2
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 24 are included; LOCF imputation was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 165 | 163 | 161
units on a scale | -0.076 (0.0369) | -0.211 (0.0373) | -0.258 (0.0371)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0005, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 2, analysis 2]; LS Mean Difference = -0.182, 95% CI 2-sided [-0.283 to -0.080]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.0091, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 2, analysis 2]; LS Mean Difference = -0.135, 95% CI 2-sided [-0.236 to -0.034]

5. Secondary Outcome: Change From Baseline in 36-item Short Form Health Survey (SF-36) Physical Functioning Domain at Week 16
Description: The Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). Norm-based scores were used in analyses, calibrated so that 50 is the average score and the standard deviation equals 10. Higher scores indicate a higher level of functioning. The physical functioning domain assesses limitations in physical activities because of health problems. A positive change from Baseline score indicates an improvement.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 16 are included; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 163 | 163 | 159
units on a scale | 1.81 (0.621) | 3.50 (0.625) | 4.23 (0.625)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0056, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 2, analysis 2]; LS Mean Difference = 2.42, 95% CI 2-sided [0.71 to 4.13]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.0504, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 2, analysis 2]; LS Mean Difference = 1.70, 95% CI 2-sided [-0.00 to 3.40]

6. Secondary Outcome: Percentage of Participants With a Modified Psoriatic Arthritis Response Criteria (PsARC) Response at Week 16
Description: Modified PsARC response is defined as improvement in at least 2 of the 4 measures, at least one of which must be tender joint count or swollen joint count, and no worsening in any of the 4 measures: • 78 tender joint count, • 76 swollen joint count, • Patient global assessment of disease activity, measured on a 100 mm visual Analog scale (VAS), where 0 mm = lowest disease activity and 100 mm = highest; • Physician global assessment of disease activity, measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest. Improvement or worsening in joint counts is defined as decrease or increase, respectively, from Baseline by ≥ 30%, and improvement or worsening in global assessments is defined as decrease or increase, respectively, from Baseline by ≥ 20 mm VAS.
Time Frame: Baseline and Week 16
Population: Full analysis set; Participants who discontinued early, or who did not have sufficient data for a definitive determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 168 | 168 | 168
percentage of participants | 29.8 | 38.7 | 46.4
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0017, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 16.7, 95% CI 2-sided [6.6 to 26.8] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 8.9, 95% CI 2-sided [-1.2 to 18.9] — [estimate comment as in outcome 3, analysis 1]

7. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 16
Description: The participant was asked to place a vertical line on a 100-mm visual analog scale on which the left-hand boundary (score = 0 mm) represents "no pain," and the right-hand boundary (score = 100 mm) represents "pain as severe as can be imagined." The distance from the mark to the left-hand boundary was recorded in millimeters.
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 165 | 163 | 159
mm | -5.7 (1.83) | -11.5 (1.85) | -13.5 (1.85)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0023, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 2, analysis 2]; LS Mean Difference = -7.9, 95% CI 2-sided [-12.9 to -2.8]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -5.8, 95% CI 2-sided [-10.8 to -0.7] — Based on an analysis of covariance (ANCOVA) model with treatment group and baseline DMARD use as factors, and the baseline value as a covariate

8. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Entheses Score (MASES) at Week 16
Description: The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) and at least 1 postbaseline value at or prior to Week 16 are included; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 95 | 100 | 108
units on a scale | -0.9 (0.30) | -1.4 (0.29) | -1.3 (0.28)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -0.4, 95% CI 2-sided [-1.2 to 0.4] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -0.5, 95% CI 2-sided [-1.3 to 0.3] — [estimate comment as in outcome 7, analysis 2]

9. Secondary Outcome: Change From Baseline in Dactylitis Severity Score at Week 16
Description: Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet will be rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline and Week 16
Population: Full analysis set. Participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) and at least 1 postbaseline value at or prior to Week 16 are included. LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 63 | 56 | 66
units on a scale | -1.4 (0.28) | -1.9 (0.31) | -1.7 (0.28)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -0.3, 95% CI 2-sided [-1.1 to 0.4] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -0.5, 95% CI 2-sided [-1.3 to 0.3] — [estimate comment as in outcome 7, analysis 2]

10. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 16
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the: • 28 tender joint count (TJC), • 28 swollen joint count (SJC), • Patient's Global Assessment of Disease Activity measured on a 10 cm visual analog scale (VAS), where 0 cm = lowest disease activity and 10 cm = highest; • Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest. The CDAI score ranges from 0 to 76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI: Remission: ≤ 2.8 Low Disease Activity: > 2.8 and ≤ 10 Moderate Disease Activity: > 10 and ≤ 22 High Disease Activity: > 22.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 16 are included. LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 158 | 160 | 158
units on a scale | -3.84 (0.929) | -8.24 (0.926) | -8.72 (0.923)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -4.88, 95% CI 2-sided [-7.41 to -2.34] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -4.39, 95% CI 2-sided [-6.92 to -1.86] — [estimate comment as in outcome 7, analysis 2]

11. Secondary Outcome: Change From Baseline in the Disease Activity Score (DAS28) at Week 16
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables: • 28 tender joint count • 28 swollen joint count, which do not include the distal interphalangeal (DIP) joints, the hip joint, or the joints below the knee; • C-reactive protein (CRP) • Patient's global assessment of disease activity. DAS28(CRP) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible level of CRP. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and Week 16
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 159 | 161 | 154
units on a scale | -0.26 (0.082) | -0.73 (0.082) | -0.79 (0.083)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -0.53, 95% CI 2-sided [-0.76 to -0.31] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -0.47, 95% CI 2-sided [-0.70 to -0.25] — [estimate comment as in outcome 7, analysis 2]

12. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 16
Description: The FACIT-Fatigue scale is a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue. A positive change from Baseline score indicates an improvement.
Time Frame: Baseline and Week 16
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 162 | 163 | 159
units on a scale | 1.55 (0.693) | 1.68 (0.696) | 3.88 (0.695)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = 2.33, 95% CI 2-sided [0.43 to 4.23] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = 0.13, 95% CI 2-sided [-1.77 to 2.03] — [estimate comment as in outcome 7, analysis 2]

13. Secondary Outcome: Change From Baseline in SF-36 Physical Function at Week 24
Description: as for outcome 5
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 163 | 163 | 161
units on a scale | 1.45 (0.671) | 3.49 (0.675) | 5.01 (0.671)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = 3.56, 95% CI 2-sided [1.72 to 5.40] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = 2.04, 95% CI 2-sided [0.21 to 3.88] — [estimate comment as in outcome 7, analysis 2]

14. Secondary Outcome: Percentage of Participants With a Modified Psoriatic Arthritis Response Criteria (PsARC) Response at Week 24
Description: Modified PsARC response is defined as improvement in at least 2 of the 4 measures, at least one of which must be tender joint count or swollen joint count, and no worsening in any of the 4 measures: •78 tender joint count, •76 swollen joint count, •Patient global assessment of disease activity, measured on a 100 mm visual Analog scale (VAS), where 0 mm = lowest disease activity and 100 mm = highest; •Physician global assessment of disease activity, measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest. Improvement or worsening in joint counts is defined as decrease or increase, respectively, from baseline by ≥ 30%, and improvement or worsening in global assessments is defined as decrease or increase, respectively, from baseline by ≥ 20 mm VAS.
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 168 | 168 | 168
percentage of participants | 18.5 | 31.0 | 42.9
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = 24.6, 95% CI 2-sided [15.2 to 34.0] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 12.4, 95% CI 2-sided [3.4 to 21.5] — [estimate comment as in outcome 3, analysis 1]

15. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 24
Description: as for outcome 7
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 165 | 163 | 162
mm | -4.2 (1.78) | -11.2 (1.79) | -14.7 (1.77)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = -10.6, 95% CI 2-sided [-15.4 to -5.7] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -7.1, 95% CI 2-sided [-12.0 to -2.2] — [estimate comment as in outcome 7, analysis 2]

16. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Entheses Score (MASES) at Week 24
Description: as for outcome 8
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) and at least 1 postbaseline value at or prior to Week 24 are included; LOCF imputation was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 96 | 100 | 110
units on a scale | -0.8 (0.31) | -1.6 (0.30) | -1.6 (0.29)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -0.8, 95% CI 2-sided [-1.6 to 0.0] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean DIfference = -0.8, 95% CI 2-sided [-1.6 to 0.1] — [estimate comment as in outcome 7, analysis 2]

17. Secondary Outcome: Change From Baseline in Dactylitis Severity Score at Week 24
Description: as for outcome 9
Time Frame: Baseline and Week 24
Population: Full analysis set. Participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) and at least 1 postbaseline value at or prior to Week 24 are included. LOCF was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 64 | 56 | 66
units on a scale | -1.3 (0.27) | -2.0 (0.30) | -1.8 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -0.5, 95% CI 2-sided [-1.2 to 0.3] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -0.7, 95% CI 2-sided [-1.5 to 0.1] — [estimate comment as in outcome 7, analysis 2]

18. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 24
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the: • 28 tender joint count (TJC), • 28 swollen joint count (SJC), • Patient's Global Assessment of Disease Activity measured on a 10 cm visual analog scale (VAS), where 0 cm = lowest disease activity and 10 cm = highest; • Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest. The CDAI score ranges from 0-76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI: Remission: ≤ 2.8; Low Disease Activity: > 2.8 and ≤ 10; Moderate Disease Activity: > 10 and ≤ 22; High Disease Activity: > 22.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 158 | 161 | 161
units on a scale | -3.14 (0.965) | -7.55 (0.958) | -9.52 (0.949)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS mean Difference = -6.38, 95% CI 2-sided [-9.00 to -3.75] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS mean Difference = -4.41, 95% CI 2-sided [-7.03 to -1.79] — [estimate comment as in outcome 7, analysis 2]

19. Secondary Outcome: Change From Baseline in the Disease Activity Score (DAS28) at Week 24
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables: • 28 tender joint count • 28 swollen joint count, which do not include the DIP joints, the hip joint, or the joints below the knee; • C-reactive protein (CRP) • Patient's global assessment of disease activity. DAS28(CRP) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible level of CRP. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 161 | 161 | 159
units on a scale | -0.20 (0.087) | -0.66 (0.087) | -0.90 (0.087)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS Mean Difference = -0.70, 95% CI 2-sided [-0.94 to -0.46] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean Difference = -0.46, 95% CI 2-sided [-0.70 to -0.22] — [estimate comment as in outcome 7, analysis 2]

20. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 24
Description: as for outcome 12
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 163 | 163 | 161
units on a scale | 1.12 (0.691) | 1.52 (0.696) | 3.33 (0.690)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; LS mean Difference = 2.21, 95% CI 2-sided [0.32 to 4.10] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; LS Mean DIfference = 0.40, 95% CI 2-sided [-1.50 to 2.29] — [estimate comment as in outcome 7, analysis 2]

21. Secondary Outcome: Percentage of Participants With MASES Improvement ≥ 20% at Week 16
Description: Percentage of participants with pre-existing enthesopathy whose MASES improved by ≥ 20% from Baseline after 16 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) are included; LOCF was used. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 98 | 103 | 114
percentage of participants | 49.0 | 56.3 | 52.6
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = 3.3, 95% CI 2-sided [-10.1 to 16.7] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 7.3, 95% CI 2-sided [-6.5 to 21.1] — [estimate comment as in outcome 3, analysis 1]

22. Secondary Outcome: Percentage of Participants With Dactylitis Improvement ≥ 1 Point at Week 16
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improved by ≥ 1 after 16 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) are included; LOCF was used. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 68 | 59 | 68
percentage of participants | 57.4 | 66.1 | 60.3
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = 2.9, 95% CI 2-sided [-13.4 to 19.3] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 7.7, 95% CI 2-sided [-9.1 to 24.6] — [estimate comment as in outcome 3, analysis 1]

23. Secondary Outcome: Percentage of Participants With Good or Moderate European League Against Rheumatism (EULAR) Response at Week 16
Description: A EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS-28 score. A Good Response is defined as an improvement (decrease) in the DAS28 of more than 1.2 compared with Baseline and attainment of a DAS28 score less than or equal to 3.2. A Moderate Response is defined as either: • an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 score of less than or equal to 5.1 or, • an improvement (decrease) in the DAS28 of more than 1.2 and attainment of a DAS28 score of greater than 3.2.
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 168 | 168 | 168
percentage of participants | 29.8 | 46.4 | 48.8
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = 19.2, 95% CI 2-sided [9.0 to 29.3] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 16.6, 95% CI 2-sided [6.4 to 26.8] — [estimate comment as in outcome 3, analysis 1]

24. Secondary Outcome: Percentage of Participants With MASES Improvement ≥ 20% at Week 24
Description: Percentage of participants with pre-existing enthesopathy whose MASES improved by ≥ 20% from Baseline after 24 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline MASES > 0 are included; LOCF was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 98 | 103 | 114
percentage of participants | 46.9 | 58.3 | 60.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = 13.2, 95% CI 2-sided [-0.1 to 26.5] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 11.3, 95% CI 2-sided [-2.4 to 25.0] — [estimate comment as in outcome 3, analysis 1]

25. Secondary Outcome: Percentage of Participants With Dactylitis Improvement ≥ 1 Point at Week 24
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improved by ≥ 1 after 24 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline dactylitis severity score > 0 are included; LOCF was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 68 | 59 | 68
percentage of participants | 60.3 | 69.5 | 69.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = 8.9, 95% CI 2-sided [-6.8 to 24.6] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 7.7, 95% CI 2-sided [-8.7 to 24.2] — [estimate comment as in outcome 3, analysis 1]

26. Secondary Outcome: Percentage of Participants With Good or Moderate EULAR Response at Week 24
Description: EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS-28 score. A Good Response is defined as an improvement (decrease) in the DAS28 of more than 1.2 compared with Baseline and attainment of a DAS28 score less than or equal to 3.2. A Moderate Response is defined as either: • an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 score of less than or equal to 5.1 or, • an improvement (decrease) in the DAS28 of more than 1.2 and attainment of a DAS28 score of greater than 3.2.
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 168 | 168 | 168
percentage of participants | 16.1 | 30.4 | 42.3
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = 26.3, 95% CI 2-sided [17.1 to 35.5] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 14.2, 95% CI 2-sided [5.4 to 23.1] — [estimate comment as in outcome 3, analysis 1]

27. Secondary Outcome: Percentage of Participants With a ACR 50 Response at Week 16
Description: Percentage of participants with an American College of Rheumatology 50% (ACR50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 50% improvement in 78 tender joint count; • ≥ 50% improvement in 76 swollen joint count; and • ≥ 50% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-Reactive Protein.
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 168 | 168 | 168
percentage of participants | 6.0 | 15.5 | 16.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = 10.3, 95% CI 2-sided [3.7 to 16.8] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 9.5, 95% CI 2-sided [3.0 to 16.0] — [estimate comment as in outcome 3, analysis 1]

28. Secondary Outcome: Percentage of Participants With an ACR 70 Response at Week 16
Description: Percentage of participants with an American College of Rheumatology 70% (ACR70) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 70% improvement in 78 tender joint count; • ≥ 70% improvement in 76 swollen joint count; and • ≥ 70% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-Reactive Protein.
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 168 | 168 | 168
percentage of participants | 1.2 | 6.0 | 4.2
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = 3.1, 95% CI 2-sided [-0.4 to 6.5] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 4.8, 95% CI 2-sided [0.8 to 8.7] — [estimate comment as in outcome 3, analysis 1]

29. Secondary Outcome: Percentage of Participants With an ACR 50 Response at Week 24
Description: as for outcome 27
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 168 | 168 | 168
percentage of participants | 4.2 | 14.3 | 19.0
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = 14.9, 95% CI 2-sided [8.3 to 21.5] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 10.1, 95% CI 2-sided [4.0 to 16.1] — [estimate comment as in outcome 3, analysis 1]

30. Secondary Outcome: Percentage of Participants With a ACR 70 Response at Week 24
Description: as for outcome 28
Time Frame: Baseline and week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 168 | 168 | 168
percentage of participants | 0.6 | 5.4 | 10.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = 9.5, 95% CI 2-sided [4.8 to 14.2] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 4.7, 95% CI 2-sided [1.2 to 8.3] — [estimate comment as in outcome 3, analysis 1]

31. Secondary Outcome: Percentage of Participants Achieving a MASES Score of Zero at Week 16
Description: Percentage of participants with pre-existing enthesopathy whose MASES improves to 0 after 16 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Week 16
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 98 | 103 | 114
percentage of participants | 15.3 | 27.2 | 22.8
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = 7.6, 95% CI 2-sided [-2.8 to 17.9] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 11.9, 95% CI 2-sided [0.8 to 23.0] — [estimate comment as in outcome 3, analysis 1]

32. Secondary Outcome: Percentage of Participants Achieving a Dactylitis Score of Zero at Week 16
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improves to zero after 16 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Week 16
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 68 | 59 | 68
percentage of participants | 39.7 | 42.4 | 38.2
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = -1.4, 95% CI 2-sided [-17.7 to 14.8] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 2.4, 95% CI 2-sided [-14.8 to 19.6] — [estimate comment as in outcome 3, analysis 1]

33. Secondary Outcome: Percentage of Participants Achieving a MASES Score of Zero at Week 24
Description: Percentage of participants with pre-existing enthesopathy whose MASES improves to 0 after 24 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Week 24
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 98 | 103 | 114
percentage of participants | 14.3 | 31.1 | 31.6
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = 17.4, 95% CI 2-sided [6.6 to 28.2] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 16.8, 95% CI 2-sided [5.6 to 27.9] — [estimate comment as in outcome 3, analysis 1]

34. Secondary Outcome: Percentage of Participants Achieving a Dactylitis Score of Zero at Week 24
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improves to zero after 24 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Week 24
Population: as for outcome 25
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 68 | 59 | 68
percentage of participants | 39.7 | 49.2 | 45.6
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; Adjusted Difference = 5.8, 95% CI 2-sided [-10.7 to 22.4] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; Adjusted Difference = 8.8, 95% CI 2-sided [-8.5 to 26.2] — [estimate comment as in outcome 3, analysis 1]

35. Secondary Outcome: Percentage of Participants With a ACR 20 Response at Week 52
Description: as for outcome 1
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population consists of all participants who were randomized or re-randomized to apremilast at any time during the study. Only those participants who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo / Apremilast 20 mg: Participants who received placebo twice daily up to Week 16 or Week 24 and were then re-randomized to receive 20 mg apremilast twice daily.
- Placebo / Apremilast 30 mg: Participants who received placebo twice daily up to Week 16 or Week 24 and were then re-randomized to receive 30 mg apremilast twice daily.
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 64 | 60 | 119 | 130
percentage of participants | 53.1 [40.2 to 65.7] | 50.0 [36.8 to 63.2] | 63.0 [53.7 to 71.7] | 54.6 [45.7 to 63.4]

36. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at Week 52
Description: as for outcome 2
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with a Baseline value and a Week 52 value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 64 | 61 | 120 | 132
units on a scale | -0.27 (0.562) | -0.29 (0.590) | -0.37 (0.479) | -0.32 (0.547)

37. Secondary Outcome: Change From Baseline in the SF-36 Physical Functioning Domain at Week 52
Description: as for outcome 5
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 64 | 61 | 120 | 130
units on a scale | 4.46 (8.877) | 4.62 (9.979) | 6.98 (9.425) | 5.69 (8.995)

38. Secondary Outcome: Percentage of Participants With a Modified PsARC Response at Week 52
Description: Modified PsARC response is defined as improvement in at least 2 of the 4 measures, at least one of which must be tender joint count or swollen joint count, and no worsening in any of the 4 measures: • 78 tender joint count, • 76 swollen joint count, • Patient global assessment of disease activity, measured on a 100 mm visual Analog scale (VAS), where 0 mm = lowest disease activity and 100 mm = highest; • Physician global assessment of disease activity, measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest. Improvement or worsening in joint counts is defined as decrease or increase, respectively, from Baseline by ≥ 30%, and improvement or worsening in global assessments is defined as decrease or increase, respectively, from Baseline by ≥ 20 mm VAS. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; only those participants who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 61 | 59 | 120 | 129
percentage of participants | 73.8 [60.9 to 84.2] | 71.2 [57.9 to 82.2] | 77.5 [69.0 to 84.6] | 73.6 [65.2 to 81.0]

39. Secondary Outcome: Change From Baseline in the Patient Assessment of Pain at Week 52
Description: as for outcome 7
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 64 | 60 | 120 | 131
mm | -20.2 (26.76) | -21.0 (25.83) | -17.8 (24.50) | -20.3 (23.37)

40. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Entheses Score (MASES) at Week 52
Description: as for outcome 8
Time Frame: Baseline and week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with a baseline value > 0 (i.e., pre-existing enthesopathy) and a Week 52 value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 36 | 36 | 69 | 89
units on a scale | -2.2 (4.03) | -1.9 (3.89) | -2.7 (2.41) | -1.9 (2.93)

41. Secondary Outcome: Change From Baseline in the Dactylitis Severity Score at Week 52
Description: as for outcome 9
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with a baseline value > 0 (i.e., pre-existing dactylitis) and a Week 52 value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 23 | 26 | 48 | 49
units on a scale | -0.8 (2.10) | -2.4 (3.58) | -2.7 (3.79) | -1.8 (3.23)

42. Secondary Outcome: Change From Baseline in the CDAI Score at Week 52
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the: • 28 tender joint count (TJC), • 28 swollen joint count (SJC), • Patient's Global Assessment of Disease Activity measured on a 10 cm visual analog scale (VAS), where 0 cm = lowest disease activity and 10 cm = highest; • Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest. The CDAI score ranges from 0-76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI: Remission: ≤ 2.8 Low Disease Activity: > 2.8 and ≤ 10 Moderate Disease Activity: > 10 and ≤ 22 High Disease Activity: > 22.
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 61 | 59 | 120 | 129
units on a scale | -15.00 (11.137) | -14.03 (14.900) | -15.41 (13.039) | -14.54 (12.009)

43. Secondary Outcome: Change From Baseline in the DAS28 at Week 52
Description: as for outcome 19
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 64 | 60 | 120 | 129
units on a scale | -1.47 (1.103) | -1.15 (1.272) | -1.40 (1.125) | -1.31 (1.114)

44. Secondary Outcome: Change From Baseline in the FACIT-Fatigue Scale Score at Week 52
Description: as for outcome 12
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 63 | 61 | 120 | 128
units on a scale | 4.33 (8.183) | 4.15 (11.712) | 4.27 (8.488) | 3.67 (9.078)

45. Secondary Outcome: Percentage of Participants With MASES Improvement ≥ 20% at Week 52
Description: Percentage of participants with pre-existing enthesopathy whose MASES improved by ≥ 20% from Baseline after 52 weeks. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; only those participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) and who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 36 | 36 | 69 | 89
percentage of participants | 69.4 [51.9 to 83.7] | 55.6 [38.1 to 72.1] | 84.1 [73.3 to 91.8] | 75.3 [65.0 to 83.8]

46. Secondary Outcome: Percentage of Participants With Dactylitis Improvement ≥ 1 Point at Week 52
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improved by ≥ 1 after 52 weeks. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; Participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) and who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 23 | 26 | 48 | 49
percentage of participants | 65.2 [42.7 to 83.6] | 73.1 [52.2 to 88.4] | 85.4 [72.2 to 93.9] | 77.6 [63.4 to 88.2]

47. Secondary Outcome: Percentage of Participants Achieving Good or Moderate EULAR Response at Week 52
Description: as for outcome 23
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Number; unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 64 | 60 | 120 | 129
percentage of participants | 82.8 | 70.0 | 75.0 | 74.4

48. Secondary Outcome: Percentage of Participants With an ACR 50 Response at Week 52
Description: Percentage of participants with an American College of Rheumatology 50% (ACR50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 50% improvement in 78 tender joint count; • ≥ 50% improvement in 76 swollen joint count; and • ≥ 50% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-Reactive Protein. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 63 | 61 | 117 | 130
percentage of participants | 25.4 [15.3 to 37.9] | 27.9 [17.1 to 40.8] | 24.8 [17.3 to 33.6] | 24.6 [17.5 to 32.9]

49. Secondary Outcome: Percentage of Participants With an ACR 70 Response at Week 52
Description: Percentage of participants with an American College of Rheumatology 70% (ACR70) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 70% improvement in 78 tender joint count; • ≥ 70% improvement in 76 swollen joint count; and • ≥ 70% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-Reactive Protein. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 62 | 61 | 117 | 130
percentage of participants | 4.8 [1.0 to 13.5] | 14.8 [7.0 to 26.2] | 15.4 [9.4 to 23.2] | 13.8 [8.4 to 21.0]

50. Secondary Outcome: Percentage of Participants Achieving a MASES Score of Zero at Week 52
Description: Percentage of participants with pre-existing enthesopathy whose MASES improves to 0 after 24 weeks. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; only those participants with a baseline value > 0 (i.e., pre-existing enthesopathy) and who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 36 | 36 | 69 | 89
percentage of participants | 33.3 [18.6 to 51.0] | 27.8 [14.2 to 45.2] | 50.7 [38.4 to 63.0] | 38.2 [28.1 to 49.1]

51. Secondary Outcome: Percentage of Participants Achieving a Dactylitis Score of Zero at Week 52
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improves to zero after 52 weeks. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Week 52
Population: as for outcome 46
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 23 | 26 | 48 | 49
percentage of participants | 52.2 [30.6 to 73.2] | 53.8 [33.4 to 73.4] | 68.8 [53.7 to 81.3] | 63.3 [48.3 to 76.6]

52. Secondary Outcome: Number of Participants With Adverse Events During the Placebo-Controlled Period
Description: A Treatment Emergent Adverse Event (TEAE) is an AE with a start date on or after the date of the first dose of Investigational Product (IP). An AE is any noxious, unintended, or untoward medical occurrence, that may appear or worsen in a participant during the course of study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) was considered an AE. A serious AE (SAE) is any untoward adverse event that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly or birth defect, or a condition that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above.
Time Frame: Week 0 to Week 16 for placebo participants who entered early escape at Week 16 and up to Week 24 for all other participants (placebo participants who remained on placebo through week 24 and participants randomized to the APR 20 mg BID or APR 30 mg BID)
Population: Safety population included all participants who were randomized and received at least one dose of IP.
Measure: Number; unit: participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 168 | 168 | 168
participants
  Treatment Emergent Adverse Events | 81 | 101 | 103
  Drug-related TEAE | 32 | 54 | 70
  Severe TEAE | 6 | 8 | 11
  Serious TEAE (SAE) | 7 | 8 | 9
  Drug-related Serious AE) | 2 | 0 | 3
  TEAE leading to drug interruption | 9 | 10 | 17
  TEAE leading to drug withdrawal | 8 | 10 | 12
  TEAE leading to drug death | 0 | 1 | 0

53. Secondary Outcome: Number of Participants With Adverse Events During the Apremilast-Exposure Period
Description: A TEAE is an AE with a start date on or after the date of the first dose of Investigational Product (IP) and no later than 28 days after the last dose of IP. An AE is any noxious, unintended, or untoward medical occurrence, that may appear or worsen in a participant during the course of study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) was considered an AE. A serious AE (SAE) is any untoward adverse event that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly or birth defect, or a condition that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above.
Time Frame: Baseline to Week 260; median total exposure to Apremilast was 170 weeks
Population: Apremilast Subjects as Treated (AAT) were those who received at least 1 dose of apremilast at any time during the study. Participants were included in the treatment group corresponding to the apremilast dosing regimen they actually received, irrespective of the treatment group to which they were randomized or re-randomized.
Measure: Number; unit: participants
Groups:
- Apremilast 20 mg (Pre-switch): Participants randomized or re-randomized to apremilast 20 mg BID and then switched to apremilast 30 mg BID (n = 87, dose switches occurring between Weeks 211 to 249). Only the TEAEs that occurred during apremilast 20 mg BID treatment were counted.
- Apremilast 20 mg/30 mg BID (Post-switch): Participants who switched from apremilast 20 mg BID to apremilast 30 mg BID. Only the TEAEs that occurred during APR 30 mg BID treatment were counted.
- Apremilast 30 mg BID: Participants who were treated with apremilast 30 mg BID throughout the study regardless of when their apremilast-exposure started (at Weeks 0, 16, or 24).
Arm/Group | Apremilast 20 mg (Pre-switch) | Apremilast 20 mg/30 mg BID (Post-switch) | Apremilast 30 mg BID
Number analyzed (Participants) | 245 | 87 | 245
participants
  Treatment Emergent Adverse Events (TEAEs) | 203 | 39 | 131
  Drug-related TEAE | 96 | 5 | 131
  Severe TEAE | 35 | 1 | 30
  Serious TEAE (SAE) | 41 | 6 | 49
  Drug-related SAE | 4 | 1 | 9
  TEAE leading to drug interruption | 47 | 3 | 49
  TEAE leading to drug withdrawal | 27 | 0 | 30
  TEAE leading to death | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: AE's are reported for the placebo-controlled phase and up to 5 years for all subjects randomized or re-randomized to apremilast at any time during the study. AEs were monitored and collected for 6 years, 4 months, 25 days excluding the end date.
Groups:
- Week 0-24: Placebo (Placebo-Controlled Phase): Subjects received placebo tablets twice daily during the placebo-controlled phase. Includes data through Week 16 for subjects who escaped early, and through Week 24 for all other subjects.
- Week 0-24: Apremilast 20 mg (Placebo- Controlled Phase): Subjects received 20 mg apremilast tablets PO BID during the 24-week placebo-controlled phase.
- Week 0-24: Apremilast 30 mg (Placebo- Controlled Phase): Subjects received 30 mg apremilast tablets PO BID during the 24-week placebo-controlled phase.
- Active Exposure up to 5 Years: Apremilast 20 mg: Subjects received 20 mg apremilast tablets BID at Week 0, and subjects initially received placebo tablets BID during the placebo controlled phase and were re-randomized and received apremilast 20 mg at Week 16 or Week 24 and continued to receive apremilast 20 mg BID for up to 4.5 years in the active treatment / long-term safety phase. Includes data which were occurring under 20 mg BID treatment.
- Active Exposure Up to 5 Years: Apremilast 20/30 mg BID: Subjects switched from apremilast 20 mg to apremilast 30 mg PO BID after identification of the optimal dose. Includes data which were occurring under 30 mg BID treatment
- Active Exposure up to 5 Years: Apremilast 30 mg BID: Subjects received 30 mg apremilast tablets BID at Week 0, and initially received placebo tablets BID during the placebo controlled phase and were re-randomized and received apremilast 30 mg at Week 16 or Week 24 and continued receiving apremilast 30 mg BID for up to 4.5 years in the active treatment / long-term safety phase.
Arm/Group | Week 0-24: Placebo (Placebo-Controlled Phase) | Week 0-24: Apremilast 20 mg (Placebo- Controlled Phase) | Week 0-24: Apremilast 30 mg (Placebo- Controlled Phase) | Active Exposure up to 5 Years: Apremilast 20 mg | Active Exposure Up to 5 Years: Apremilast 20/30 mg BID | Active Exposure up to 5 Years: Apremilast 30 mg BID
Serious Adverse Events (participants affected / at risk) | 7/168 | 8/168 | 9/168 | 41/245 | 6/87 | 49/245
Other Adverse Events (participants affected / at risk) | 43/168 | 69/168 | 80/168 | 150/245 | 17/87 | 169/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Week 0-24: Placebo (Placebo-Controlled Phase) (N=168) | Week 0-24: Apremilast 20 mg (Placebo- Controlled Phase) (N=168) | Week 0-24: Apremilast 30 mg (Placebo- Controlled Phase) (N=168) | Active Exposure up to 5 Years: Apremilast 20 mg (N=245) | Active Exposure Up to 5 Years: Apremilast 20/30 mg BID (N=87) | Active Exposure up to 5 Years: Apremilast 30 mg BID (N=245)
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 2
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Incision site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 2
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Wound infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Yersinia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Borderline personality disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 3 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 1
Thinking abnormal (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Week 0-24: Placebo (Placebo-Controlled Phase) (N=168) | Week 0-24: Apremilast 20 mg (Placebo- Controlled Phase) (N=168) | Week 0-24: Apremilast 30 mg (Placebo- Controlled Phase) (N=168) | Active Exposure up to 5 Years: Apremilast 20 mg (N=245) | Active Exposure Up to 5 Years: Apremilast 20/30 mg BID (N=87) | Active Exposure up to 5 Years: Apremilast 30 mg BID (N=245)
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 8 | 11 | 1 | 13
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3 | 7 | 5 | 0 | 15
Diarrhoea (Gastrointestinal disorders) | 4 | 20 | 32 | 33 | 1 | 51
Dyspepsia (Gastrointestinal disorders) | 4 | 4 | 6 | 8 | 1 | 14
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 5 | 10 | 1 | 19
Nausea (Gastrointestinal disorders) | 11 | 16 | 32 | 30 | 0 | 41
Bronchitis (Infections and infestations) | 2 | 2 | 0 | 17 | 3 | 19
Gastroenteritis (Infections and infestations) | 0 | 3 | 3 | 16 | 0 | 11
Nasopharyngitis (Infections and infestations) | 5 | 7 | 8 | 30 | 3 | 31
Sinusitis (Infections and infestations) | 4 | 4 | 4 | 21 | 2 | 21
Upper respiratory tract infection (Infections and infestations) | 6 | 10 | 7 | 41 | 3 | 36
Urinary tract infection (Infections and infestations) | 3 | 3 | 2 | 10 | 3 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 12 | 0 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 14 | 0 | 13
Headache (Nervous system disorders) | 8 | 17 | 18 | 31 | 2 | 34
Anxiety (Psychiatric disorders) | 1 | 2 | 0 | 7 | 0 | 14
Depression (Psychiatric disorders) | 1 | 4 | 1 | 17 | 1 | 10
Insomnia (Psychiatric disorders) | 3 | 2 | 3 | 13 | 0 | 9
Hypertension (Vascular disorders) | 2 | 6 | 2 | 20 | 4 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.